CLINICAL TRIAL: NCT00124410
Title: A Pilot Study to Determine the Prevalence of Osteoporosis in Patients With Advanced Prostate Cancer Treated With Hormonal Manipulation
Brief Title: Study to Determine the Prevalence of Osteoporosis in Patients With Advanced Prostate Cancer Treated With Hormonal Manipulation
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NA-15-0001
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2011-12

CONDITIONS: Prostate Cancer; Osteoporosis
Keywords: prostate cancer; androgen suppression therapy (hormone therapy); osteoporosis
MeSH Terms: conditions — Prostatic Neoplasms; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Osteoporosis, or thinning of the bones is a common disorder which can cause significant morbidity in terms of pain and fracture. One of the causes of osteoporosis is a low or absent testosterone level. Prostate cancer is the second most common malignancy in males with an increasing incidence. The mainstay of advanced prostate cancer treatment is hormonal manipulation (surgery or medications) in order to lower testosterone levels as testosterone stimulates cancer cells. Despite the known links both between osteoporosis, low testosterone, and prostate cancer, little data is available on how common osteoporosis is among men with advanced prostate cancer treated with hormonal manipulation. Since prostate cancer affects so many men and the indications for early hormonal manipulation are expanding, it is important to determine the prevalence of osteoporosis in these males.

DETAILED DESCRIPTION:
INTRODUCTION - Osteoporosis is a common disorder with many predisposing factors including hypogonadism from a variety of causes. Prostate cancer is the second most common malignancy in men. The standard treatment for men with advanced prostate cancer is hormonal manipulation in order to decrease testosterone levels which renders a man hypogonadal. There is an increasing body of literature that suggests men with prostate cancer treated with hormonal manipulation develop osteoporosis and associated complications more commonly than aged matched controls. With the increasing incidence of prostate cancer and the increasing indications with hormonal therapy use in advanced prostate cancer, osteoporosis in these men is a major health concern.Hormonal manipulation in order to obtain castrate levels of testosterone can be achieved with bilateral orchiectomy, Luteinizing Hormone Releasing Hormone agonists (LHRHA) and steroidal antiandrogens combined with mini doses of estrogen based therapy. Nonsteroidal antiandrogens are also used in the management of advanced prostate cancer however, on their own, are not enough to suppress testosterone. The data on exactly how common and severe a problem osteoporosis is in men treated with different forms of hormonal manipulation is sparse and because of the lack of data, there is currently no accepted standard of care in the investigation and management of osteoporosis in these men. The researchers propose to start with a pilot study to first determine the prevalence of osteoporosis in 6 different populations of men with advanced prostate cancer, (1) newly diagnosed, (2) treated with orchiectomy, (3) treated with an LHRHA, (4) treated with steroidal antiandrogen therapy, (5) treated with nonsteroidal antiandrogen based therapy, (6) treated with complete androgen blockade (LHRHA plus a nonsteroidal antiandrogen).

OBJECTIVES - To determine, in the above populations, the bone mineral density as measured by Dual Energy X-ray Absorptiometry (DEXA) of the lumbar spine, proximal hip (total hip, femoral neck and trochanter), and non-dominant distal radius, to document biochemical markers of bone turnover, to document vertebral fractures and body height, to document other aspects of body composition including adipose tissue and muscle mass as measured by whole body composition densitometry, and to document other potential confounding factors predisposing prostate cancer patients to osteoporosis.

STUDY DESIGN - This primarily will be a descriptive, exploratory study describing the prevalence of osteoporosis in each of the 6 groups defined above. The diagnosis of osteoporosis will be based on bone densitometry studies. There are accepted densitometric criteria for the assessment of normal and abnormal bone mass. The criteria were largely developed in postmenopausal Caucasian women but reference values are also available for Caucasian, Black and Hispanic men. Normal bone density is described as a T-score less than -1. T-scores between -1 and -2.5 are indicative of osteopenia, and T-scores of less than -2.5 are indicative of osteoporosis. The prevalence of osteoporosis (T value less than 2.5) in each of the groups will be reported. Information on biochemical markers of bone turnover, vertebral fractures, and other risk factors will also be described.

PATIENT SELECTION - Patients with biopsy proven advanced prostate cancer, no known prior clinical or radiographic history of osteoporosis, minimum of 1 year of hormonal therapy in arms 2, 3, 4, 5 and 6, and an ability and willingness to give informed consent. Exclusion criteria - Patients with known bone disorders other than metastatic disease such as hyperparathyroidism, Paget's disease, renal osteodystrophy, and documented osteomalacia as well as osteoporosis, patients who have received a bisphosphonate, systemic fluoride, pharmacological doses of calcium (less than 1500 mg/day) or Vitamin D (less than 1000 IU/day), or calcitonin, patients with known abnormal thyroid function, and patients with marked renal impairment (creatinine less than 2.0 X normal).

MANAGEMENT OF PATIENTS - This will be an outpatient study. All patients will initially be assessed by a research nurse and/or physician at the Cross Cancer Institute with a prostate cancer specific history, blood and urine tests. Patients will be referred to a single endocrinologist for a more detailed osteoporosis history and physical exam. On the same day, they will have a densitometry study, whole body composition study, and plain radiographs taken. Patients will then be seen at the Cross Cancer Institute to discuss their results. Should a diagnosis of osteoporosis be made, a letter indicating this will be sent to the patient's family physician.

ENDPOINTS - The primary endpoint will be bone mineral density. Osteoporosis will be diagnosed if the T value is less than -2.5. The secondary endpoints will be - biochemical markers of bone turnover, vertebral fractures, vertebral body height, body composition of fat, body composition of adipose tissue.

DATA ANALYSIS - The data will be entered into a computerized database. Descriptive statistics will be tabulated for all 5 arms being studied with respect to demographic variables, baseline characteristics, and test results.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients, on hormone therapy

Exclusion Criteria:

* No prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2000-01; Primary Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Venner, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada